CLINICAL TRIAL: NCT01257789
Title: Structured Bariatric Fellowship Programme Moelholm Private Hospital - Denmark. Learning Laparoscopic RY - Gastric Bypass One Way to do it
Brief Title: Eliminating Learning Curve Related Morbidity in Fast Track Laparoscopic Roux-en-Y Gastric Bypass
Status: Completed | Type: Observational
Sponsor: Private Hospital Moelholm (Other)
Responsible Party: Thorbjorn Sommer, Private Hospital Moelholm
Other Study IDs: PHM-GB learning study
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-02

CONDITIONS: Postoperative Complications; Operative Time; Surgical Volume
Keywords: laparoscopic gastric bypass; learning curve; complications; operative time
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- gastric bypass patients: Consecutive series of 300 patients undergoing laparoscopic gastric bypass
  Interventions: Procedure: laparoscopic gastric bypass

INTERVENTIONS:
Procedure: laparoscopic gastric bypass — laparoscopic gastric bypass

SUMMARY:
Background: Laparoscopic Roux en Y gastric bypass (LRYGB) is associated with a significant learning curve. We report the results of a systematic training programme from a high volume bariatric center measuring the outcome by comparing the results with data from a consecutive series of 1000 fast track LRYGB.

Method: Using a stepwise training programme the RY gastric bypass operation was divided into an upper and lower procedure and subdivided into 11 well defined steps. A laparoscopic surgeon without experience in upper GI surgery was mentored by an experienced bariatric surgeon. During 6 months full time fellowship 300 operations were performed.

Results: The trainee surgeon performed 61 upper procedures, and 121 lower procedures in which the mentor surgeon did the other part of the operation. In 110 patients the trainee performed both procedures. Two percent had peri-operative complications compared to 1% of 1000 patients. All were repaired and had an uneventful recovery. Two percent had postoperative complications < 30 days compared to 2.8% in the clinic. In the trainees series there were no leaks compared to 1% in 1000 patients. Operative time was 56/55/70 min for operation 0-100/100-200/200-300 compared with an average of 47 minutes registered in the clinic. Concerning time to discharge there was no difference between patients operated by the trainee and the standard of the clinic.

Conclusion: Using a systematic training program in laparoscopic RY gastric bypass surgery eliminates morbidity of the learning curve without affecting the volume.

ELIGIBILITY:
Inclusion Criteria:

patients undergoing laparoscopic gastric bypass

Exclusion Criteria:

* super obesity
* male patients

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 consequtive patients already sceduled for laparoscopic gastric bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
complication rate
  data of all postoperative complications untill 4 months post OP were collected

CONTACTS AND LOCATIONS:
Locations (1):
- Private Hospital Moelholm, Vejle, Denmark